CLINICAL TRIAL: NCT05345197
Title: Emicizumab in Patients With Acquired Hemophilia A: Multicenter, Single-arm, Open-label Clinical Trial
Brief Title: Emicizumab in Patients With Acquired Hemophilia A
Acronym: AHAEmi
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Kruse-Jarres, Professor, School of Medicine: Hematology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00013920
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-06

CONDITIONS: Acquired Hemophilia A
Keywords: Acquire Hemophilia A; emicizumab; AHA
MeSH Terms: conditions — Factor 8 deficiency, acquired | interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental-treatment (Experimental): Treatment with emicizumab
  Interventions: Drug: emicizumab

INTERVENTIONS:
Drug: emicizumab — This study design uses emicizumab as a prophylaxis treatment to prevent bleeding for all participants, bypassing agents (with the exception of aPCC) and treatment of concomitant diseases will be given as clinically indicated. All eligible subjects with AHA will receive the same study medication consisting of: two loading doses of the emicizumab on day 1 and 2 followed by once weekly subcutaneous emicizumab injections. Immunosuppressive therapy (IST) will be given concurrently as per investigator discretion.
  Other Names: Hemlibra (R)

SUMMARY:
This is a phase II multicenter open-label, single-arm prospective study to evaluate the efficacy of prophylactic emicizumab administered on a scheduled basis to prevent bleeds in patients with acquired hemophilia A (AHA).

DETAILED DESCRIPTION:
Patients with AHA who are eligible will receive two loading doses of the study drug, emicizumab (6mg/kg on day 1 and 3 mg/kg on day 2) followed by once weekly subcutaneous emicizumab (1.5 mg/kg). Immunosuppression will be given concurrently as per investigator discretion. The primary endpoint (bleed rate) will be assessed after 12 weeks on study drug. If partial remission of the AHA has not been achieved, an additional 12 weeks of study drug may be given. A historical cohort and a study conducted in parallel in Germany (NCT04188639) will serve as control groups for evaluation of secondary endpoints provided the study cohort are comparable.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent/Assent Form
* Age ≥18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Diagnosis of AHA based on a reduced FVIII activity (<50 %) and positive FVIII inhibitor (>0.6 BU/ml) at screening (local laboratory)
* Current bleeding due to AHA at the time of screening
* Plan to be adherent to emicizumab prophylaxis during the study
* For women of childbearing potential who meet the following criteria:
* Refrain from heterosexual intercourse or use contraceptive methods that result in a failure rate of <1% per year during the study period A woman with ≥ 12 continuous months of amenorrhea with no identified cause other than menopause and has not undergone surgical sterilization (removal of ovaries and/or uterus). use of combined oral or injected hormonal contraceptive, bilateral tubal ligation, male sterilization, hormone- releasing intrauterine devices, and copper intrauterine devices.

Exclusion Criteria:

* Congenital hemophilia A
* Treatment with aPCC within the last 24 hours before first study treatment or planned treatment with aPCC during the course of the study
* Known positive lupus anticoagulant at the time of screening
* Severe uncontrolled infection at the time of screening
* Signs of active disseminated intravascular coagulation at the time of screening -
* Emicizumab ⎯ AHA Emi Version 1.0 20
* Current treatment for thromboembolic disease or signs of current thromboembolic disease at time of screening
* Patients who are at high risk for TMA (e.g., have a previous medical or family history of TMA), in the investigator's judgment
* Known severe congenital or acquired thrombophilia
* Life expectancy <3 months at the time of screening
* Other conditions that substantially increase risk of bleeding or thrombosis by the discretion of the investigator
* Contraindications according to the Investigator's Brochure of emicizumab
* Current treatment with emicizumab at time of screening
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection by the discretion of the investigator
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose additional risk, or would, in the opinion of the local investigator, preclude the patient's safe participation in and completion of the study
* Addiction or other diseases that preclude the patient from appropriately assessing the nature and scope as well as possible consequences of the clinical study by the discretion of the investigator
* Pregnant or breast-feeding women
* Would refuse treatment with blood or blood products, if necessary.
* Subject is in custody by order of an authority or a court of law
* Treatment with any of the following:
* An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration before Study Day 1
* A non-hemophilia-related investigational drug within the last 30 days or 5 half-lives- before Study Day 1, whichever is longer
* An investigational drug concurrently
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Meassure | 12 weeks
  Number of clinically significant bleeds after 12 weeks of study drug (emicizumab)

SECONDARY OUTCOMES:
Incidence and severity of adverse events | duration of entire study
  Incidence and severity of adverse events, including thromboembolic events, thrombotic microangiopathy in the 12 weeks after starting emicizumab treatment; mortality and cause of death in the 24 weeks after starting emicizumab treatment.
Days of treatment with additional hemostatic agent | 12 weeks
  Days of treatment with and total dose of bypassing agents (recombinant factor VIIa, activated prothrombin complex concentrate) or recombinant porcine factor VIII (susoctocag alfa) or other factor VIII concentrates; specifics (drug, amount and timing) of IST started during the 12 weeks of emicizumab prophylaxis
Remission Rate | 1 to 24 weeks
  Number of patients achieving partial remission (PR) and complete remission (CR) over 12 and 24 weeks after starting emicizumab prophylaxis
Hospitalizations | 12 weeks
  Days in hospital during week 12 of emicizumab treatment
Total dose of additional hemostatic agent | 12 weeks
  Total dose of bypassing agents (recombinant factor VIIa, activated prothrombin complex concentrate) or recombinant porcine factor VIII (susoctocag alfa) or other factor VIII concentrates; specifics (drug, amount and timing) of IST started during the 12 weeks of emicizumab prophylaxis

OTHER OUTCOMES:
Comparison of historic GTH-AH 01/2020 cohort/ Number of clinically significant bleeds | 12 to 24 weeks
  Number of clinically significant bleeds in the 12 weeks of emicizumab treatment or until achieving partial remission (PR) of AHA, whatever occurs first Incidence and severity of adverse events, thromboembolic events, thrombotic microangiopathy, in 12 weeks of treatment and mortality after 24 weeks Bleeding-free survival until week 12 after starting treatment
Comparison to a parallel German study cohort/ Number of clinically significant bleeds | 12 to 24 weeks
  Number of clinically significant bleeds per patient-week until death or week 12 after starting emicizumab treatment, whatever occurs first Incidence and severity of adverse events, thromboembolic events, in the 12 weeks of emicizumab treatment and mortality after 24 weeks Bleeding-free survival until week 12 of emicizumab treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kruse-Jarres, MD, MPH, Principal Investigator — University of Washington
Locations (16):
- United States (16):
  - UCSD Hemophilia and Thrombosis Treatment Center, San Diego, California
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center, Inc., Indianapolis, Indiana
  - Tulane University, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn Blood Disorders Program, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - University of Vermont Medical Center, Burlington, Vermont
  - UVA Comprehensive Cancer Center, Charlottesville, Virginia
  - Washington Center for Bleeding Disorders, Seattle, Washington
  - Versiti Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared with the research group of the parallel European study (NCT04188639). Data will be shared at the end of the study for analysis for a period of 2 years.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared with the research group of the parallel European study (NCT04188639) at the end of the study and will be available for 2 years.
Access Criteria: Only researchers of this or the parallel trial (NCT04188639) will have access to this data.

REFERENCES:
- [Background] Franchini M, Gandini G, Di Paolantonio T, Mariani G. Acquired hemophilia A: a concise review. Am J Hematol. 2005 Sep;80(1):55-63. doi: 10.1002/ajh.20390. PMID 16138334
- [Background] Kruse-Jarres R, Kempton CL, Baudo F, Collins PW, Knoebl P, Leissinger CA, Tiede A, Kessler CM. Acquired hemophilia A: Updated review of evidence and treatment guidance. Am J Hematol. 2017 Jul;92(7):695-705. doi: 10.1002/ajh.24777. Epub 2017 Jun 5. PMID 28470674
- [Background] Kessler CM, Knobl P. Acquired haemophilia: an overview for clinical practice. Eur J Haematol. 2015 Dec;95 Suppl 81:36-44. doi: 10.1111/ejh.12689. PMID 26679396
- [Background] Tiede A, Amano K, Ma A, Arkhammar P, El Fegoun SB, Rosholm A, Seremetis S, Baudo F. The use of recombinant activated factor VII in patients with acquired haemophilia. Blood Rev. 2015 Jun;29 Suppl 1:S19-25. doi: 10.1016/S0268-960X(15)30004-7. PMID 26073365
- [Background] Sallah S. Treatment of acquired haemophilia with factor eight inhibitor bypassing activity. Haemophilia. 2004 Mar;10(2):169-73. doi: 10.1046/j.1365-2516.2003.00856.x. PMID 14962206
- [Background] Kruse-Jarres R, St-Louis J, Greist A, Shapiro A, Smith H, Chowdary P, Drebes A, Gomperts E, Bourgeois C, Mo M, Novack A, Farin H, Ewenstein B. Efficacy and safety of OBI-1, an antihaemophilic factor VIII (recombinant), porcine sequence, in subjects with acquired haemophilia A. Haemophilia. 2015 Mar;21(2):162-170. doi: 10.1111/hae.12627. Epub 2015 Jan 27. PMID 25623166
- [Background] Tiede A, Scharf RE, Dobbelstein C, Werwitzke S. Management of acquired haemophilia A. Hamostaseologie. 2015;35(4):311-8. doi: 10.5482/HAMO-14-11-0064. Epub 2015 Jan 7. PMID 25564260
- [Background] Tiede A, Klamroth R, Scharf RE, Trappe RU, Holstein K, Huth-Kuhne A, Gottstein S, Geisen U, Schenk J, Scholz U, Schilling K, Neumeister P, Miesbach W, Manner D, Greil R, von Auer C, Krause M, Leimkuhler K, Kalus U, Blumtritt JM, Werwitzke S, Budde E, Koch A, Knobl P. Prognostic factors for remission of and survival in acquired hemophilia A (AHA): results from the GTH-AH 01/2010 study. Blood. 2015 Feb 12;125(7):1091-7. doi: 10.1182/blood-2014-07-587089. Epub 2014 Dec 18. PMID 25525118
- [Background] Knoebl P, Thaler J, Jilma P, Quehenberger P, Gleixner K, Sperr WR. Emicizumab for the treatment of acquired hemophilia A. Blood. 2021 Jan 21;137(3):410-419. doi: 10.1182/blood.2020006315. PMID 32766881
- [Background] Al-Banaa K, Alhillan A, Hawa F, Mahmood R, Zaki A, El Abdallah M, Zimmerman J, Musa F. Emicizumab Use in Treatment of Acquired Hemophilia A: A Case Report. Am J Case Rep. 2019 Jul 18;20:1046-1048. doi: 10.12659/AJCR.916783. PMID 31318850
- [Background] Mohnle P, Pekrul I, Spannagl M, Sturm A, Singh D, Dechant C. Emicizumab in the Treatment of Acquired Haemophilia: A Case Report. Transfus Med Hemother. 2019 Apr;46(2):121-123. doi: 10.1159/000497287. Epub 2019 Mar 15. PMID 31191199
- [Background] Muto A, Yoshihashi K, Takeda M, Kitazawa T, Soeda T, Igawa T, Sampei Z, Kuramochi T, Sakamoto A, Haraya K, Adachi K, Kawabe Y, Nogami K, Shima M, Hattori K. Anti-factor IXa/X bispecific antibody ACE910 prevents joint bleeds in a long-term primate model of acquired hemophilia A. Blood. 2014 Nov 13;124(20):3165-71. doi: 10.1182/blood-2014-07-585737. Epub 2014 Oct 1. PMID 25274508
- [Background] Rodriguez-Merchan EC, Valentino LA. Emicizumab: Review of the literature and critical appraisal. Haemophilia. 2019 Jan;25(1):11-20. doi: 10.1111/hae.13641. Epub 2018 Nov 15. PMID 30431213
- [Background] Levy GG, Asikanius E, Kuebler P, Benchikh El Fegoun S, Esbjerg S, Seremetis S. Safety analysis of rFVIIa with emicizumab dosing in congenital hemophilia A with inhibitors: Experience from the HAVEN clinical program. J Thromb Haemost. 2019 Sep;17(9):1470-1477. doi: 10.1111/jth.14491. Epub 2019 Jun 17. PMID 31124272
- [Background] Pipe SW, Shima M, Lehle M, Shapiro A, Chebon S, Fukutake K, Key NS, Portron A, Schmitt C, Podolak-Dawidziak M, Selak Bienz N, Hermans C, Campinha-Bacote A, Kiialainen A, Peerlinck K, Levy GG, Jimenez-Yuste V. Efficacy, safety, and pharmacokinetics of emicizumab prophylaxis given every 4 weeks in people with haemophilia A (HAVEN 4): a multicentre, open-label, non-randomised phase 3 study. Lancet Haematol. 2019 Jun;6(6):e295-e305. doi: 10.1016/S2352-3026(19)30054-7. Epub 2019 Apr 16. PMID 31003963
- [Background] Mahlangu J, Oldenburg J, Paz-Priel I, Negrier C, Niggli M, Mancuso ME, Schmitt C, Jimenez-Yuste V, Kempton C, Dhalluin C, Callaghan MU, Bujan W, Shima M, Adamkewicz JI, Asikanius E, Levy GG, Kruse-Jarres R. Emicizumab Prophylaxis in Patients Who Have Hemophilia A without Inhibitors. N Engl J Med. 2018 Aug 30;379(9):811-822. doi: 10.1056/NEJMoa1803550. PMID 30157389
- [Background] Langer AL, Etra A, Aledort L. Evaluating the safety of emicizumab in patients with hemophilia A. Expert Opin Drug Saf. 2018 Dec;17(12):1233-1237. doi: 10.1080/14740338.2019.1551356. Epub 2018 Nov 28. PMID 30462521
- [Background] Young G, Callaghan M, Dunn A, Kruse-Jarres R, Pipe S. Emicizumab for hemophilia A with factor VIII inhibitors. Expert Rev Hematol. 2018 Nov;11(11):835-846. doi: 10.1080/17474086.2018.1531701. Epub 2018 Oct 10. PMID 30278802
- [Background] Mahlangu J. Emicizumab for the prevention of bleeds in hemophilia A. Expert Opin Biol Ther. 2019 Aug;19(8):753-761. doi: 10.1080/14712598.2019.1626370. Epub 2019 Jun 13. PMID 31150297
- [Background] Shima M, Hanabusa H, Taki M, Matsushita T, Sato T, Fukutake K, Fukazawa N, Yoneyama K, Yoshida H, Nogami K. Factor VIII-Mimetic Function of Humanized Bispecific Antibody in Hemophilia A. N Engl J Med. 2016 May 26;374(21):2044-53. doi: 10.1056/NEJMoa1511769. PMID 27223146
- [Background] Collins PW, Liesner R, Makris M, Talks K, Chowdary P, Chalmers E, Hall G, Riddell A, Percy CL, Hay CR, Hart DP. Treatment of bleeding episodes in haemophilia A complicated by a factor VIII inhibitor in patients receiving Emicizumab. Interim guidance from UKHCDO Inhibitor Working Party and Executive Committee. Haemophilia. 2018 May;24(3):344-347. doi: 10.1111/hae.13495. PMID 30070072
- [Background] Oldenburg J, Mahlangu JN, Kim B, Schmitt C, Callaghan MU, Young G, Santagostino E, Kruse-Jarres R, Negrier C, Kessler C, Valente N, Asikanius E, Levy GG, Windyga J, Shima M. Emicizumab Prophylaxis in Hemophilia A with Inhibitors. N Engl J Med. 2017 Aug 31;377(9):809-818. doi: 10.1056/NEJMoa1703068. Epub 2017 Jul 10. PMID 28691557
- [Background] Takeyama M, Nogami K, Matsumoto T, Noguchi-Sasaki M, Kitazawa T, Shima M. An anti-factor IXa/factor X bispecific antibody, emicizumab, improves ex vivo coagulant potentials in plasma from patients with acquired hemophilia A. J Thromb Haemost. 2020 Apr;18(4):825-833. doi: 10.1111/jth.14746. Epub 2020 Feb 26. PMID 31984625
- [Background] Devarajan P, Chen Z. Autoimmune effector memory T cells: the bad and the good. Immunol Res. 2013 Dec;57(1-3):12-22. doi: 10.1007/s12026-013-8448-1. PMID 24203440
- [Background] Tiede A, Hofbauer CJ, Werwitzke S, Knobl P, Gottstein S, Scharf RE, Heinz J, Gross J, Holstein K, Dobbelstein C, Scheiflinger F, Koch A, Reipert BM. Anti-factor VIII IgA as a potential marker of poor prognosis in acquired hemophilia A: results from the GTH-AH 01/2010 study. Blood. 2016 May 12;127(19):2289-97. doi: 10.1182/blood-2015-09-672774. Epub 2016 Feb 24. PMID 26912467
- [Background] Mongini PK, Paul WE, Metcalf ES. T cell regulation of immunoglobulin class expression in the antibody response to trinitrophenyl-ficoll. Evidence for T cell enhancement of the immunoglobulin class switch. J Exp Med. 1982 Mar 1;155(3):884-902. doi: 10.1084/jem.155.3.884. PMID 6977611
- [Background] Pavlova A, Zeitler H, Scharrer I, Brackmann HH, Oldenburg J. HLA genotype in patients with acquired haemophilia A. Haemophilia. 2010 May;16(102):107-12. doi: 10.1111/j.1365-2516.2008.01976.x. PMID 20536993
- [Background] Holling TM, Schooten E, van Den Elsen PJ. Function and regulation of MHC class II molecules in T-lymphocytes: of mice and men. Hum Immunol. 2004 Apr;65(4):282-90. doi: 10.1016/j.humimm.2004.01.005. PMID 15120183